CLINICAL TRIAL: NCT02738034
Title: Cogmed Training Effect in Hypertensive Patients With Cognitive Impairment: a Randomized Clinical Trial
Brief Title: Cogmed Training Effect in Hypertensive Patients With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Regina Silva Paradela, PhD student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CogDoc2016
Record Dates: First submitted 2016-03-23; First posted 2016-04-14 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2020-11

CONDITIONS: Hypertension
Keywords: Hypertension; Cognition; Computerized Training; Cogmed
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Adaptive training group (Experimental): The intervention group will be composed of hypertensive participants with cognitive decline that will be submitted to the training program (Cogmed) for approximately 10 weeks. Across training, task difficulty was adjusted as a function of individual performance.
  Interventions: Other: Cogmed
- Active control Group (Active Comparator): In the control group, hypertensive patient will be submitted to a set of online games available on the internet and previously determined. In this way, the control group will receive the same motivation, as well as will be engaged in computerized activities, in the same way as the experimental group. The difference is that these varied games do not provide any type of intense and adaptive training, at the same time as they do not stimulate any specific cognitive function.
  Interventions: Other: Cogmed

INTERVENTIONS:
Other: Cogmed — The Cogmed is computer software designed to train visuospatial and audio-verbal working memory, and other functions associated with working memory: attention, focus and impulsiveness. It has three versions adapted to different age groups: Cogmed for younger children, about 4-7 years, which are not yet so familiar with numbers and letters; Cogmed for children over 7 years and adolescents; and Cogmed for youth and adults over 18 years. In this study we will use the version for youth and adults over 18 years.

SUMMARY:
Systemic arterial hypertension is a disease with high prevalence in several countries, including Brazil. Many studies have correlated hypertension with accelerated loss of cognitive function, especially executive functions. There is some evidence that working memory (WM) is compromised in these populations. However, some computerized training has been developed to rehabilitate the WM, and among them the investigators highlight the Cogmed. Thus, the aim of this study is to evaluate the effects of Cogmed training in the performance of WM and attention of hypertensive patients, as well as the impact of training in the structure and brain function.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders, of any ethnicity
* Signing the consent form
* Access to computer with internet at home
* Inexperienced to computerized cognitive training
* Hypertensive pre-diagnosed
* Basic schooling of four years
* Cognitive impairment

Exclusion Criteria:

* Marked functional limitation
* Cognitive limitation or serious communication
* Severe neurological and psychiatric diseases
* Stroke history, head trauma or substance abuse

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Working memory score | 10 weeks
  Backward Digits Test / Letter-Number Sequencing (WAIS-III): total score (sum of right answers)

SECONDARY OUTCOMES:
Brain function | 10 weeks
  Functional magnetic resonance
Executive functions score | 10 weeks
  Stroop test, Wisconsin Card Sorting Test, Frontal Assessment Battery and Controlled Oral Word Association Test
Verbal memory score | 10 weeks
  Stories of Wechsler Memory Scale Revised - WMS R
Visual memory score | 10 weeks
  Rey complex figure

OTHER OUTCOMES:
Medication adherence score | 10 weeks
  Short version of Morinsk Questionnaire
Quality of life score | 10 weeks
  Whoqol
Perceived Stress score | 10 weeks
  PSS14
Anxiety and Depression symptoms score | 10 weeks
  BAI and BDI questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Silva Paradela, São Paulo, São Paulo, Brazil